CLINICAL TRIAL: NCT07002450
Title: Left Atrial Imaging Prior to Cardioversion: Leveraging Computed Tomography to Rule Out Thrombus in The Emergency Department (LA CLOTTED)
Acronym: LA CLOTTED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20240752-01T
Record Dates: First submitted 2025-05-08; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation (AF); Atrial Flutter
Keywords: Cardiac computed tomography angiography; Cardioversion; Atrial flutter; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Patients in the control arm will be treated according to current standard of care as determined by the primary treating emergency department physician and may vary by institution and physician. Treatment in the standard of care group may include a rate control strategy with or without a planned cardioversion after 3 weeks of anticoagulation, deferring management for outpatient evaluation, request for TEE-facilitated cardioversion in the ED, or specialist consultation for further management or admission to hospital.
  Interventions: Other: Standard of care management
- CCT-facilitated cardioversion arm (Experimental): Patients in this arm will undergo cardiac computed tomography angiography (CCT) to evaluate for a left atrial/left atrial appendage (LA) thrombus. If the CCT shows no LA thrombus then the emergency department physician will be able to perform electrical and/or chemical cardioversion at their discretion. If the CCT shows a LA thrombus then cardioversion will be contraindicated and further management will be at the discretion of the treating physician.
  Interventions: Diagnostic Test: Cardiac computed tomography angiography

INTERVENTIONS:
Diagnostic Test: Cardiac computed tomography angiography — Patients will undergo CCT according to the following protocol. A non-contrast enhanced prospective ECG-triggered image will be acquired followed by a contrast-enhanced prospective ECG-triggered image using a tri-phasic contrast protocol. Delayed CT images 60 seconds after the initial contrast-enhanced CT scan will be obtained. Cardiac CT image interpretation will be performed according to routine clinical practices in a pragmatic fashion. The LA will be assessed for filling defects and characterized based upon attenuation values. If LA thrombus cannot be excluded, filling defects will be assessed on the delay images. Increases in attenuation would be consistent with pseudo-thrombus from 'slow flow' and 'incomplete opacification'. Areas where attenuation does not change significantly (persistent filling defect) will be diagnosed as thrombus. If the CCT shows no LA thrombus then the ED physician will be able to perform electrical and/or chemical cardioversion at their discretion.
  Arms: CCT-facilitated cardioversion arm
Other: Standard of care management — Patients in the standard of care arm may undergo any combination of the following management strategies in the emergency department (ED) at the discretion of their treating physician:
  1. Transesophageal echocardiogram (TEE) facilitated cardioversion; 2. Rate control; 3. Consultation with inpatient cardiac specialist for assessment/management and consideration of hospital admission; 4. cardioversion after 3 weeks of anticoagulation; and/or 5. Outpatient referral to cardiac specialist or general practitioner for further management.
  Arms: Standard of Care

SUMMARY:
The goal of this randomized clinical trial is to learn whether patients with symptomatic atrial fibrillation or atrial flutter (AF) who require heart imaging to rule out a blood clot before cardioversion would benefit from cardiac computed tomography angiography (CCT) in the emergency department (ED) compared to current standard of care management.

This will be a multicenter trial evaluating whether CCT-facilitated cardioversion in the ED reduces hospital admission, reduces repeat presentations to hospital and improves patient quality of life compared to the current standard of care.

Participants will undergo CCT-facilitated cardioversion or be treated according to current standard of care while in the ED and complete quality of life questionnaires in the ED and follow-up at 30 days.

DETAILED DESCRIPTION:
Atrial fibrillation and atrial flutter (AF) are the most common cardiac arrhythmias worldwide resulting in frequent visits to the emergency department (ED). Some patients can undergo chemical or electrical cardioversion to restore their heart back to a sinus rhythm. However, if a patient is not on blood thinners and the duration of AF is prolonged then blood clots may form in the heart increasing the risk of stroke after cardioversion. Therefore, some patients must undergo heart imaging to rule out any blood clots before cardioversion is considered safe. Transesophageal echocardiography (TEE) is commonly used to rule out blood clots, but it is not readily available in all EDs often resulting in hospital admission to facilitate this test or deferring cardioversion until 3 weeks of blood thinners have been completed.

Cardiac computed tomography angiography (CCT) is a more readily available alternative to TEE that can be done rapidly in the ED. CCT has excellent sensitivity and specificity compared to TEE for identifying cardiac thrombus. If there is no thrombus detected on the CCT then patients could be immediately cardioverted to sinus rhythm thus avoiding an unnecessary hospital admission and reducing the symptom burden associated with remaining in AF.

This study is a multicenter randomized trial that will evaluate the effectiveness of using CCT facilitated cardioversion in the ED compared to current standard of care management.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old; and
2. Primary symptomatic AF without a reversible underlying cause (e.g. sepsis, pneumonia, pulmonary embolism, hyperthyroidism)
3. LA imaging required before cardioversion according to local clinical practice guidelines

Exclusion Criteria:

1. Patients with an indication for emergency cardioversion (e.g. hemodynamic instability (systolic blood pressure<90mmHg or signs of shock), cardiac ischemia (ongoing severe chest pain or marked ST depression on ECG >2mm), or pulmonary edema (significant dyspnea, crackles, or hypoxia)); or
2. Contraindication to CCT (renal insufficiency (eGFR< 45ml/min/1.73m2), allergy to intravenous contrast agents, pregnancy (contraindications to radiation exposure), or inability to perform 20-second breath-hold)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Primary composite outcome | Randomization to 30 days
  Using a hierarchical win ratio:
  1. All-cause death
  2. Stroke, transient ischemic attack, or systemic embolism
  3. Admission to hospital for a cardiac reason (ex. heart failure, syncope, palpitations/arrhythmia, angina or acute coronary syndrome)
  4. Number of repeat presentations to hospital for a cardiac reason (ex. heart failure, syncope, palpitations/arrhythmia, angina or acute coronary syndrome)
  5. Improvement in AF Effect On Quality-Of-Life Questionnaire (AFEQT) quality of life greater than or equal to 5 points
  6. Presence of sinus rhythm at 30 days

SECONDARY OUTCOMES:
Composite secondary outcome | Randomization to 30 days
  Using a hierarchical win ratio:
  1. All-cause death
  2. Stroke, transient ischemic attack, or systemic embolism
  3. Admission to hospital for a cardiac reason (ex. heart failure, syncope, palpitations/arrhythmia, angina or acute coronary syndrome)
  4. Number of repeat presentations to hospital for a cardiac reason (ex. heart failure, syncope, palpitations/arrhythmia, angina or acute coronary syndrome)
  5. Improvement in AF Effect On Quality-Of-Life Questionnaire (AFEQT) quality of life greater than or equal to 5 points
Composite objective outcomes | Randomization to 30 days
  Using a hierarchical win ratio:
  1. All-cause death
  2. Stroke, transient ischemic attack, or systemic embolism
  3. Admission to hospital for a cardiac reason (ex. heart failure, syncope, palpitations/arrhythmia, angina or acute coronary syndrome)
  4. Number of repeat presentations to hospital for a cardiac reason (ex. heart failure, syncope, palpitations/arrhythmia, angina or acute coronary syndrome)
All-cause death | Randomization to 30 days
  Death from any cause
Cardiovascular death | Randomization to 30 days
  Death due to a cardiovascular cause
Stroke, transient ischemic attack, or systemic embolism | Randomization to 30 days
  Stroke is defined as a central nervous system infarction of the brain, spinal cord, or retina in a vascular distribution based on pathologic, imaging, or clinical evidence with symptoms persisting for ≥24 hours or until death.
  Transient ischemic attack is defined as a transient episode of neurologic dysfunction due to focal brain, spinal cord, or retinal ischemia without acute infarction or tissue injury.
  Systemic embolism is defined as an abrupt vascular insufficiency associated with clinical or radiologic evidence of arterial occlusion in the absence of other likely mechanisms.
Hospital admission for a cardiac reason | Randomization to 30 days
  Hospitalization due to a cardiac reason such as heart failure, syncope, palpitations/arrhythmia, angina or acute coronary syndrome
Repeat presentation to the emergency department | Randomization to 30 days
  Repeat presentation to the emergency department due to a cardiac reason such as heart failure, syncope, palpitations/arrhythmia, angina or acute coronary syndrome
AFEQT quality of life | Randomization to 30 days
  Change in AF Effect On Quality-Of-Life Questionnaire (AFEQT) quality of life The AFEQT is a 20-item, self-administered instrument that quantifies symptoms, daily activities, treatment concern, and treatment satisfaction. Scores are transformed to a range from 0-100, in which higher scores reflect better health status.
SF-36 quality of life | Randomization to 30 days
  Change in 36-Item Short Form Health Survey (SF-36) quality of life. The SF-36 questionnaire consists of eight scales yielding two summary measures: physical and mental health. The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items). Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Bleeding | Randomization to 30 days
  Bleeding events as defined by the Bleeding Academic Research Consortium
Admission to hospital for acute kidney injury | Randomization to 30 days
  Definition of acute kidney injury according to the Kidney Disease Improving Global Outcomes:
  * Increase in SCr by ≥ 0.3 mg/dl (≥ 26.5 µmol/l) within 48 hours; or
  * Increase in SCr to ≥ 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or
  * Urine volume <0.5 ml/kg/h for 6 hours
Length of stay in the emergency department | From time of arrival until time of discharge or admission (approximately 3 hours)
  Length of stay in emergency department in minutes, from time of arrival to time of discharge or admission
Normal sinus rhythm | At the time of patient disposition (approximately 3 hours after arrival)
  Being in normal sinus rhythm at the time of emergency department disposition (discharge or admission). Heart rhythm will be determined by electrocardiography.

OTHER OUTCOMES:
Cost effectiveness | Emergency department presentation to 30 days
  Cost effectiveness between CCT strategy and standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Chow, MD PhD FRCPC FACC FESC FA, Principal Investigator — Ottawa Heart Institute Research Corporation; Mehrdad Golian, MD MSC FRCPC, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- The Ottawa Hospital Civic Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The study data, protocol, SAP, ICF, and CSR will be made available at study completion/publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study completion
Access Criteria: The above will be made publicly available.